CLINICAL TRIAL: NCT00268762
Title: A Pilot Study To Determine The Safety Of Argatroban Injection In Combination With Tissue Plasmingen Activator (TPA) In Patients With Acute Ischemic Stroke
Brief Title: Argatroban Stroke Treatment - A Pilot Safety Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Andrew Barreto, Assistant Professor - Neurology, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Argatroban+TPA 02-121B; P50NS44227 project #2 (Other Grant/Funding Number: P50NS44227); P50NS044227 (NIH)
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Ischemic Stroke
Keywords: stroke; thrombin inhibition; thrombolysis; bleeding; outcome
MeSH Terms: conditions — Ischemic Stroke; Stroke; Hemorrhage | interventions — argatroban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Argatroban IV Infusion 1 mcg/kg/min for 48 hours
  Interventions: Drug: argatroban

INTERVENTIONS:
Drug: argatroban — Argatroban IV Infusion at 1mcg/kg/min for 48 hours.

SUMMARY:
Is the combination of low doses of argatroban in combination with rt-PA safe, and does it increase recanalization in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
All patients with acute ischemic stroke who qualify for IV rt-PA under accepted guidelines, and who have an occluded middle cerebral artery documented on TCD, receive standard dose IV rt-PA and a bolus and 48 hour infusion of argatroban aimed at prolonging the aPTT 1.75 X baseline. Follow up CT scanning and TCD every 30 minutes for 2 hours and then daily will determine the incidence of hemorrhage, recanalization and reocclusion, and serial neurological exam will determine the clinical outcome. For patients without temporal windows, a baseline CT-Angiogram (CTA) demonstrating arterial occlusion can also be enrolled. In those patients, a follow-up CTA (24-36 hours) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke symptoms with onset ≤ 3 hours*.

  * *or<4.5 hours according to local standard of care. Symptoms must be distinguished from another ischemic event such as syncope, seizure, migraine, and hypoglycemia. If the patient reports awakening with the event, the time of onset should be considered as last time the patient (or a witness to the patient's condition) considered herself/himself normal.
* 18-85 years of age.
* A clot causing complete or partial occlusion (TIBI 0, 1, 2, or 3) via TCD in any one of the following areas: distal iternal carotid artery (ICA), Meddle cerebral artery (MCA - M1 or M2), posterior cerebral arteral (ICA - P1 or P2), distal vertebral or basilar occlusions. TCD must be abnormal prior to the start of Argatroban. For patients without temporal windows (or in centers without emergent access to TCD), an abnormal CTA is required for enrollment (TIMI 0 or 1).
* Females of childbearing potential must have a negative serum pregnancy test prior administration of argatroban.
* Signed informed consent by the patient or the patient's legal representative.
* Meet criteria for rt-PA therapy.

Exclusion Criteria:

* Evidence of intracranial hemorrhage on baseline CT scan or non-vascular cause of neurologic deficit.
* National institute health stroke scale (NIHSS) Level of Consciousness score ≥2.
* Baseline (immediately pre-Argatroban) NIHSS ≤ 5 or patient with rapidly resolving deficit or rapidly improving symptoms consistent with TPA.
* Baseline NIHSS ≥15 for right hemisphere strokes and ≥20 for left hemisphere strokes.
* Pre-existing disability with modified rankin scale (mRS) ≥ 2.
* CT scan findings of hypoattenuation of the x-ray signal (hypodensity)involving ≥ 1/2 of the MCA territory.
* Any evidence of clinically significant bleeding, or known coagulopathy.
* Patients currently on warfarin, with an elevated INR ≥ 1.5.
* Patients currently or within previous 48 hrs. on heparin with an elevated aPTT greater than the upper limit of normal.
* Heparin flush required for an IV line. Line flushes with saline only.
* History of ICH or significant bleeding episode within the 3 months before study enrollment.
* Major surgery or serious trauma within the last 6 weeks.
* Patients who have had an arterial puncture at a non-compressible site, biopsy of parenchymal organ, or lumbar puncture within the last 2 weeks.
* Previous stroke, myocardial infarction, post myocardial infarction pericarditis, intracranial surgery, or significant head trauma within 3 months of baseline.
* Uncontrolled hypertension.
* Alcohol and/or substance abuse that would increase the risk of hemorrhage in the opinion of the investigator.
* Surgical intervention anticipated within the next 7 days.
* Hepatic dysfunction, defined by liver function tests greater than 3 times upper limit of normal at baseline, specifically serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamic-pyruvic transaminase (SGPT).
* Abnormal blood glucose
* History of primary or metastatic brain tumor.
* Severe mental deficit prior to onset of stroke such as organic brain disorder, schizophrenia, etc.
* Concurrent severe neurologic disorder, such as seizure at onset of stroke or uncontrolled seizure disorder that complicates diagnosis of acute ischemic stroke.
* Current platelet count< 100,000/mm3.
* Life expectancy <3 months in the opinion of the investigator.
* Need to be on concomitant (i.e, during the Argatroban infusion) anticoagulants other than Argatroban, including any form of heparin, unfractionated heparin (UFH), low molecular weight heparin (LMWH), defibrinogenating agent, dextran, other direct thrombin inhibitors or thrombolytic agents, glycoprotein llb/llla (GPIIb/IIIa) or warfarin.(Caveat: If these anticoagulants can be deferred for 48 hours, then they can be included).
* Participated in investigational study within 30 days before the first dose of study medication.
* Hypersensitivity to Argatroban or its agents

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2003-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D. Barreto, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (6):
- United States (6):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Tulane University, New Orleans, Louisiana
  - University of Texas-Southwestern Dallas, Dallas, Texas
  - Memorial Hermann Hospital-Medical Center, Houston, Texas
  - Memorial Hermann Southwest Hospital, Houston, Texas

REFERENCES:
- [Result] Sugg RM, Pary JK, Uchino K, Baraniuk S, Shaltoni HM, Gonzales NR, Mikulik R, Garami Z, Shaw SG, Matherne DE, Moye LA, Alexandrov AV, Grotta JC. Argatroban tPA stroke study: study design and results in the first treated cohort. Arch Neurol. 2006 Aug;63(8):1057-62. doi: 10.1001/archneur.63.8.1057. PMID 16908730
- [Result] Barreto AD, Alexandrov AV, Lyden P, Lee J, Martin-Schild S, Shen L, Wu TC, Sisson A, Pandurengan R, Chen Z, Rahbar MH, Balucani C, Barlinn K, Sugg RM, Garami Z, Tsivgoulis G, Gonzales NR, Savitz SI, Mikulik R, Demchuk AM, Grotta JC. The argatroban and tissue-type plasminogen activator stroke study: final results of a pilot safety study. Stroke. 2012 Mar;43(3):770-5. doi: 10.1161/STROKEAHA.111.625574. Epub 2012 Jan 5. PMID 22223235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first enrollment: May 6, 2003 Date of last enrollment: August 20, 2010 All patients enrolled through hospital emergency departments
Groups:
- Intervention: Argatroban IV bolus 100 mcg/kg bolus, followed by Argatroban IV Infusion 1 mcg/kg/min for 48 hours. Dose adjusted for target partial thromboplastin time (PTT) of 1.75 times the patient's baseline.
Period: Overall Study
Arm/Group | Intervention
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Argatroban IV bolus 100 mcg/kg bolus, followed by Argatroban IV Infusion 1 mcg/kg/min for 48 hours. Dose adjusted for target PTT of 1.75 times the patient's baseline.
Arm/Group | Intervention
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic and Radiographic Intracerebral Hemorrhage
Description: Significant intracerebral hemorrhage as defined by either:
  1. Symptomatic intracerebral hemorrhage or
  2. Parenchymal hematoma type 2.
Time Frame: Within 7 days of enrollment
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Intervention
Number analyzed (Participants) | 65
percentage of patients | 6.2 [1.7 to 15.0]

2. Secondary Outcome: Arterial Complete Recanalization at 2 Hours Post tPA Bolus
Description: Complete Recanalization as measured by either transcranial Doppler Ultrasound at 2 hours post tPA bolus.
Time Frame: 2 hours complete recanalization post tPA bolus
Measure: Number; unit: percent of patients
Arm/Group | Intervention
Number analyzed (Participants) | 47
percent of patients | 40

3. Secondary Outcome: Arterial Complete Recanalization at 24 Hours Post tPA Bolus
Description: Complete recanalization at 24 hours post tPA bolus as measured by either transcranial Doppler ultrasound or CT-Angiography.
Time Frame: 24 hours from tPA bolus
Measure: Number; unit: percent of patients
Arm/Group | Intervention
Number analyzed (Participants) | 60
percent of patients | 63

ADVERSE EVENTS:
Time Frame: 90 days during the study period
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 21/65
Other Adverse Events (participants affected / at risk) | 55/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=65)
Death (General disorders) | 7 (7) — Death that occured by any of the following causes: (brain herniation or respiratory failure)
Stroke progression or neurological worsening (Nervous system disorders) | 5 (5)
Significant intracerebral hemorrhage (Nervous system disorders) | 4 (4) — Significant intracerebral hemorrhage defined as either: 1. Symptomatic intracerebral hemorrhage or 2. Parenchymal Hematoma - type 2
Cerebral edema (Nervous system disorders) | 4 (4)
Pneumonia/respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cardiac arrest (Cardiac disorders) | 3 (3)
Asymptomatic ICH (Nervous system disorders) | 2 (2)
Significant laboratory abnormality (Blood and lymphatic system disorders) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=65)
Nausea with or without Emesis (Gastrointestinal disorders) | 3 (3)
Chest Pain (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 3 (3) — This includes one patient with "Low Blood Pressure"
Tachycardia (Cardiac disorders) | 7 (7)
Patent Foramen Ovale (Cardiac disorders) | 1 (1) — New diagnosis of patent foramen ovale.
Aortic valve vegetation (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Hypothermia (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 3 (3)
Laboratory abnormalities - Chemistries (General disorders) | 10 (14) — Elevated: Creatinine Kinase/troponin=6; Liver Function Tests=2; blood urea nitrogen (BUN)=1; myoglobin=1 ; Bilirubin=1; Ketones=1; Serum Creatinine=1; Hypoglycemia=1
New diagnosis of diabetes mellitus (Endocrine disorders) | 2 (2)
Oliguria (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Urinary Analysis laboratory abnormality (Renal and urinary disorders) | 3 (3) — Leuko-Uria = 1 & Hematuria = 2
Anemia/decrease in hemoglobin and hematocrit level (Blood and lymphatic system disorders) | 4 (5)
Asymptomatic Intracranial Hemorhhage (Nervous system disorders) | 13 (13)
Fever (Infections and infestations) | 17 (17)
Urinary Tract Infection (Infections and infestations) | 19 (19)
Pneumonia (Infections and infestations) | 3 (3)
Minimally displaced fracture of base of fifth metacarpal (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hand swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Agitation/lethargic/somnolent (Nervous system disorders) | 2 (2)
Stroke progression (Nervous system disorders) | 2 (2)
Neuro-worsening (Nervous system disorders) | 3 (3)
Exacerbation of uterine prolapse (General disorders) | 1 (1)
Oral thrush (General disorders) | 1 (1)
Excessive sleepness (Psychiatric disorders) | 1 (1)
Self extubation (General disorders) | 1 (1)
Visual hallucination (Psychiatric disorders) | 1 (1)
Restless (Psychiatric disorders) | 1 (1)
Right lung mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coughing/gagging (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Both lung with rales (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Slight angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Laboratory Abnormalities - Electrolytes (General disorders) | 13 (19) — Hypokalemia=5; Hyperkalemia=2; Hyponatremia=3; Hypernatremia=2; Hypocalcemia=3 Hypomagnesia=1; Hypophosphatemia=2; Electrolyte disorder not-specified=1
Laboratory Abnormalities - Elevated PTT >100 seconds (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Possible selection bias and investigators unblinded to treatment. In addition, although 60/65 patients had 24 hour recanalization data, only 47 were available at 2 hours.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No